CLINICAL TRIAL: NCT05772039
Title: Minimally Invasive Treatment Approach for Early Childhood Caries Using Silver Diammine Fluoride and Sodium Fluoride With Functionalized Tricalcium Phosphate and Their Effects on Oral Health Related Quality of Life: A Pragmatic Randomized Control Trial
Brief Title: Treatment of Early Childhood Caries Using Silver Diammine Fluoride and Sodium Fluoride Tricalciumphosphate and the Effects on Oral Health Related Quality of Life
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: 3M ESPE (Industry); SDI Limited (Unknown)
Responsible Party: Principal Investigator, ANAS IMRAN ARSHAD, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USM/JEPeM/20010069
Record Dates: First submitted 2023-02-13; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Early Childhood Caries; Dental Caries in Children; Dental Caries Extending Into Dentin; Dental Caries; Behavior, Child; Quality of Life
Keywords: SDF; NaF-fTCP; child behavior; pain experience; Wong-Baker Faces Pain rating scale; oral health-related quality of life; caries arrest; caries prevention; silver diammine fluoride; minimal intervention dentistry; Functionalized tricalcium phosphate; Sodium fluoride
MeSH Terms: conditions — Dental Caries; Child Behavior | interventions — silver diamine fluoride; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Topical application of 38% Silver Diammine Fluoride Solution at Baseline (Active Comparator): * SDF is known for its corrosive nature therefore a plastic container or dappen dish will be used.
  * 1 drop (0.05 ml) will be dispensed on a plastic container.
  * 1 drop (2.24 F-ion mg/dose) SDF treats up to 5 tooth surfaces.
  * Ultrafine microbrushes will be used to apply varnish.
  Interventions: Drug: Topical application of 38% Silver Diammine Fluoride Solution
- Topical application of 38% Silver Diammine Fluoride Solution at 6 months (Active Comparator): * SDF is known for its corrosive nature therefore a plastic container or dappen dish will be used.
  * 1 drop (0.05 ml) will be dispensed on a plastic container.
  * 1 drop (2.24 F-ion mg/dose) SDF treats up to 5 tooth surfaces.
  * Ultrafine microbrushes will be used to apply varnish.
  Interventions: Drug: Topical application of 38% Silver Diammine Fluoride Solution
- Topical application of 38% Silver Diammine Fluoride Solution at 12 months (Active Comparator): * SDF is known for its corrosive nature therefore a plastic container or dappen dish will be used.
  * 1 drop (0.05 ml) will be dispensed on a plastic container.
  * 1 drop (2.24 F-ion mg/dose) SDF treats up to 5 tooth surfaces.
  * Ultrafine microbrushes will be used to apply varnish.
  Interventions: Drug: Topical application of 38% Silver Diammine Fluoride Solution
- Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish at baseline (Experimental): * 0.25 ml of the solution will be used which contains 12.5 mg of fluoride.
  * Thin layer will be applied with sweeping horizontal brush strokes to all teeth present.
  Interventions: Drug: Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish
- Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish at 6 months (Experimental): * 0.25 ml of the solution will be used which contains 12.5 mg of fluoride.
  * Thin layer will be applied with sweeping horizontal brush strokes to all teeth present.
  Interventions: Drug: Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish
- Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish at 12 months (Experimental): * 0.25 ml of the solution will be used which contains 12.5 mg of fluoride.
  * Thin layer will be applied with sweeping horizontal brush strokes to all teeth present.
  Interventions: Drug: Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish

INTERVENTIONS:
Drug: Topical application of 38% Silver Diammine Fluoride Solution — * Application of petroleum jelly on lips and around the mouth for prevention of temporary silver tattoo.
  * Before SDF application, the affected area will be thoroughly dried and isolated using the cotton rolls or dri-angle.
  * Isolation throughout the procedure and following three minutes is considered most desirable.
  * The varnish should be allowed to be in place for 60 seconds. This is the most critical step in the process. Applied varnish will be dried with gentle flow of compressed air.
  * SDF will be applied with a microbrush to all carious lesions and to all pits and fissures on posterior (molar) teeth for 60 seconds.
  * To avoid gingival or mucosal irritation, contact of varnish with any oral tissue other than affected area will be avoided.
  * If the application time is shorter due to unforeseen reasons reapplication will be considered.
  Other Names: Riva Star; 38% Silver Diammine fluoride; SDF; Advanatge Arrest; Saforide
  Arms: Topical application of 38% Silver Diammine Fluoride Solution at 12 months; Topical application of 38% Silver Diammine Fluoride Solution at 6 months; Topical application of 38% Silver Diammine Fluoride Solution at Baseline
Drug: Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish — * According to manufacturer, Clinpro® White Varnish can be applied to tooth surfaces where plaque is present. A prophylaxis is not required.
  * The applicator brush provided along is used to thoroughly mix the varnish inside the single-unit dose pack, since components of all sodium fluoride varnishes are separate during storage.
  * Excessive contact with soft tissue should be avoided.
  * Only enough varnish to form a thin coating on the desired treatment area should be used.
  * After application, patient should be instructed to close their mouth to set the varnish.
  * Rinsing or suctioning immediately after application is not recommended.
  * The operator might appreciate the formation of a thin coating on the teeth and the patient should be informed that they may feel a thin coating when rubbing the treated area with their tongue.
  Other Names: ClinPro White varnish; Sodium fluoride with functionalized tricalcium phosphate; NaF-fTCP
  Arms: Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish at 12 months; Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish at 6 months; Topical application of 5% Sodium Fluoride with functional Tricalcium phosphate Varnish at baseline

SUMMARY:
There is still a need for the assessment of different minimal intervention strategies and treatments focusing on the prevention and arrest of carious lesions of primary molars The evidence-based clinical practice guideline on non-restorative treatments for cavitated carious lesions advocate the use of silver diammine fluoride biannually for high caries risk patients

DETAILED DESCRIPTION:
Although SDF has been proven to be highly effective in carious lesion arrest and prevention, the staining effect, metallic taste due to silver content and the minimal mucosal irritation have been noted as primary cause of disinterest among clinicians in the use of this material.

The use of NaF-fTCP as a caries preventive material has not been studied widely. The importance of oral hygiene education and diet modification to achieve an effective caries control has been widely discussed. The off-label use of NaF-fTCP as a caries arresting agent has not been studied on primary dentition. There is a dearth of evidence regarding the effectiveness of NaF-fTCP towards caries arrest and prevention in pragmatic settings.

A comparison between the SDF and NaF-fTCP application on the cavitated carious primary molars and their effect on the oral health-related quality of life of the children has not been published in the literature.

ELIGIBILITY:
Inclusion criteria:

Children will be invited to participate in the trial if they fulfil the entire selection criteria as described below:

* 4 to 6 years-of-age
* Identification of one or more carious primary molars without involvement of the pulp confirmed by bitewing radiographs
* Up to three teeth per each participant will be selected for intervention
* Has normal salivary flow rate
* Does not consume medications regularly for any medical condition
* Has not or will not receive any fluoride therapy or relevant dental therapy from other dental sources within the last six months

Exclusion criteria:

Children will be excluded from the trial if they fulfil any of the following criteria:

* Presence of any pain, ulceration, fistula/sinus or an abscess
* Premature hypermobility of carious teeth which can be potentially included in the study
* History of allergy to any product containing silver compounds
* Siblings of the participants will not be allowed to participate to ensure any chance of ECOHIS duplication.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Caries prevalence | Baseline
  Calculated by the frequency of participants having decayed, missing, filled surfaces of dentition
Frequency distribution of caries risk | Baseline
  Calculated using Caries Risk Assessment questionnaire, which is denoted as low, moderate or high
Mean score of oral health impact | Baseline
  Calculated using Urdu-Early Childhood Oral Health Impact Scale form, the answer for each item is on a 5-point scale. The sum score of answers to the 13 questions can range from 0-52. The impact of oral health on life activities is predicted to be greater with a higher score in the summation which denotes a poorer quality of life.
Patient behaviour towards dental treatment | Baseline
  Calculated using Frankl behaviour rating scale four category which are: definitely negative, negative, positive, definitely positive
Mean score of pain experience | Baseline
  Calculated using Wong Baker Faces Scale on a range of facial expression where 0 denotes no pain, 2, 4, 6 ,8 and 10 denotes the most painful experience
Mean value of caries experience | Baseline
  Calculated by summation of number of decayed, missing and filled surfaces of dentition
Extent of selected cavitated carious lesion using ICDAS | Baseline
  Coded according to ICDAS-2 scoring system code 3: Moderate enamel breakdown, code 4: Moderate underlying dentinal shadow 5: extensive carious lesion extending to dentin without pulpal involvement
Extent of selected cavitated carious lesion using FOTI | Baseline
  Coded using Fiber optic transillumination device corresponding to ICDAS code 3- code 5
Changes in the mean score of oral health impact | 6 months
  Calculated using Urdu-Early Childhood Oral Health Impact Scale form, the answer for each item is on a 5-point scale. The sum score of answers to the 13 questions can range from 0-52. The impact of oral health on life activities is predicted to be greater with a higher score in the summation which denotes a poorer quality of life.
Changes in the mean score of patient behaviour towards dental treatment | 6 months
  Calculated using Frankl behaviour rating scale four category which are: definitely negative, negative, positive, definitely positive
Changes in the mean score of pain experience | 6 months
  Calculated using Wong Baker Faces Scale on a range of facial expression where 0 denotes no pain, 2, 4, 6 ,8 and 10 denotes the most painful experience
Changes in the mean value of caries experience | 6 months
  Calculated by summation of number of decayed, missing and filled surfaces of dentition
Extent of selected cavitated carious lesion using ICDAS | 6 months
  Coded according to ICDAS-2 scoring system code 3: Moderate enamel breakdown, code 4: Moderate underlying dentinal shadow 5: extensive carious lesion extending to dentin without pulpal involvement
Extent of selected cavitated carious lesion using FOTI | 6 months
  Coded using Fiber optic transillumination device corresponding to ICDAS code 3- code 5
Changes in the mean score of oral health impact | 12 months
  Calculated using Urdu-Early Childhood Oral Health Impact Scale form, the answer for each item is on a 5-point scale. The sum score of answers to the 13 questions can range from 0-52. The impact of oral health on life activities is predicted to be greater with a higher score in the summation which denotes a poorer quality of life.
Changes in the mean score of patient behaviour towards dental treatment | 12 months
  Calculated using Frankl behaviour rating scale four category which are: definitely negative, negative, positive, definitely positive
Changes in the mean score of pain experience | 12 months
  Calculated using Wong Baker Faces Scale on a range of facial expression where 0 denotes no pain, 2, 4, 6 ,8 and 10 denotes the most painful experience
Changes in the mean value of caries experience | 12 months
  Calculated by summation of number of decayed, missing and filled surfaces of dentition
Extent of selected cavitated carious lesion using ICDAS | 12 months
  Coded according to ICDAS-2 scoring system code 3: Moderate enamel breakdown, code 4: Moderate underlying dentinal shadow 5: extensive carious lesion extending to dentin without pulpal involvement
Extent of selected cavitated carious lesion using FOTI | 12 months
  Coded using Fiber optic transillumination device corresponding to ICDAS code 3- code 5

SECONDARY OUTCOMES:
Number of participants reporting adverse events | Baseline
  The frequency of participants reporting fluoride or silver toxicity
Percentage of dropouts | 6 months
  Frequency of participants which either withdraw and do not consent for follow up
Number of participants reporting adverse events | 6 months
  The frequency of participants reporting fluoride or silver toxicity
Percentage of dropouts | 12 months
  Frequency of participants which either withdraw and do not consent for follow up
Number of participants reporting adverse events | 12 months
  The frequency of participants reporting fluoride or silver toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anas Imran Arshad, MSc., BDS, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Crescent Montessori School, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient data will only be used for knowledge transfer and personal information of each patient will be kept private and confidential. After performing data analysis and report writing the collected patient data will be securely transferred to hospital archives which are not accessible without proper identification and authorization. Data from the archives will be automatically erased after two years.

DOCUMENTS (1):
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT05772039/ICF_000.pdf